CLINICAL TRIAL: NCT05959317
Title: Effect of 6-weeks Pilates Exercise Versus Neural Dynamic Mobilization on Pain, Flexibility and Quantity of Life in Patients With Sciatica.
Brief Title: Effects of Pilates Exercises and Neural Dynamic Mobilization in Sciatica Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Maria Iqbal
Record Dates: First submitted 2023-03-31; First posted 2023-07-25 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Sciatica
Keywords: Neurodynamic Mobilization
MeSH Terms: conditions — Sciatica | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Exercises (Other): Pilates exercises will be perform for 15-30 minutes for one session 3 days a week for 6-weeks than after 6 week reassess the QOL, pain and flexibility.
  Interventions: Other: Pilates Exercises
- Neural dynamic mobilization (Other): Neural dynamic mobilization will be perform for 15-30 minutes for one session 3 days a week for 6-weeks after 6 weeks reassess the QOL, pain and flexibility.
  Interventions: Other: Neural dynamic mobilization

INTERVENTIONS:
Other: Pilates Exercises — Pilates exercises will be perform for 15-30 minutes for one session 3 days a week for 6-weeks than after 6 week reassess the QOL, pain and flexibility.
  Arms: Pilates Exercises
Other: Neural dynamic mobilization — Neural dynamic mobilization will be perform for 15-30 minutes for one session 3 days a week for 6-weeks after 6 weeks reassess the QOL, pain and flexibility.
  Arms: Neural dynamic mobilization

SUMMARY:
The main purpose of the study is to find the effects of Pilates exercises and neural mobilization techniques on pain, flexibility and quality of life in sciatica patients. It will be a randomized controlled trial in which participants selected through non probability convenience sampling, to evaluate the effect of 6-week Pilates exercises versus neural dynamic mobilization techniques on pain, flexibility and quality of life in sciatica patients. Patients aged range from 18 to 65 years. The data will be collected from Service Hospital Lahore. Patients will have diagnosed with sciatica low back pain radiating down hip to knee, numbness, paresthesia and with positive SLR will include in this study whereas patients with considerable musculoskeletal deformity, previous hip, knee and ankle surgery and foot ulceration will be excluded from study .The participants will be randomly allocated to one of the two groups. Group A will perform Pilates mats exercises 30 minutes, two times a week and the Group B will perform neural dynamic mobilization for 15 minutes, two times a week, for 6-weeks respectively. Pain will be assessed by using BPFS, flexibility with Canadian sit to reach test and QOL with SF-36 questionnaire. SPSS software will be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* o Participants age ranged from 18 to 65 years old

  * Both genders.
  * History of nonspecific low back
  * lower extremity symptoms such as tingling, dull aches or burning sensation.

Exclusion Criteria:

* o Significant musculoskeletal deformity such as fracture, amputation.

  * Prior history of knee or back surgery
  * Lower extremity arthritis that limits standing and any inflammatory disease
  * History of cardiovascular issues such as angina, MI
  * Symptomatic postural hypotension
  * Foot ulceration.
  * Skin problems such as rashes etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Back pain functional questionnaire to access pain | Changes from baseline Back Pain Function Scale (BPFS) at 1.5 months
  The Back Pain Function Scale (BPFS) of Stratford et al Overview: Stratford et al developed the Back Pain Function Scale (BPFS) to evaluation functional ability in patients with back pain. The authors are from McMaster University Appalachian Physical Therapy (Georgia) and Virginia Commonwealth University. Interpretation: • minimum score: 0 • maximum score: 60 • maximum adjusted score: 1 (100%) • The higher the score the greater the patient's functional ability. Total Score (Adjusted) Interpretation: 0 (0%) unable to perform any activity 60 (100%) no difficulty in any activity Performance
Sit and reach test for flexibility | Changes from baseline Sit and reach test at 1.5 months
  Sit and Reach Test The objective of this test is to monitor the development of the athlete's lower back and hamstring flexibility. Required resources to undertake this test you will require: 'Sit & reach' table or a bench with a ruler for Assistant. This test is suitable for active individuals but not for those where the test would be contraindicated.
SF-36 questionnaire to access quality of life | Changes from baseline Short Form 36 Health Survey Questionnaire (SF-36) at 1.5 months
  The Short Form 36 Health Survey Questionnaire (SF-36) is used to indicate the health status of particular populations, to help with service planning and to measure the impact of clinical and social interventions.
  To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Iqbal, DPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Service Hospital Lahore, Lahore, Punjab Province
  - Service Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vartak HS, Rajapurkar R, Palekar T, Saini S, Khisty A. A comparative study between neural mobilisation techniques versus nerve flossing technique in patients with acute sciatica. International Journal of Basic and Applied Research. 2019;9(3):909-22.